CLINICAL TRIAL: NCT02077894
Title: Whole Exome and Whole Genome Sequencing for Genotyping of Inherited and Congenital Eye Conditions
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140064; 14-EI-0064
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12-12

CONDITIONS: Genetic Eye Disease
Keywords: Whole Genome Sequencing; Genetic Eye Disease; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected participants: Participants with an eye disease.
- Unaffected family members: Unaffected family members.

SUMMARY:
Objective: The objective of this study is to identify genetic causes of inherited eye conditions through whole exome or whole genome sequencing (referred to as exome sequencing and genome sequencing in the remainder of the document). This includes identifying mutations in known genes or novel genes for recognized conditions, as well as identifying mutations in novel genes for previously uncharacterized genetic conditions involving the eye.

Study Population: We plan to recruit 1,685 participants, to include both participants with an eye condition under study and unaffected family members. Ideally unaffected family members will be parents of an affected participant.

Design: Participants will be self-referred or referred by an outside clinician. They will preferably be evaluated at the National Institutes of Health (NIH), but the option to participate offsite will be offered. Participants evaluated onsite will be recruited through other pre-existing NIH protocols, such as the National Eye Institute (NEI) Screening protocol (08-EI-0102), the NEI Ocular Natural History protocol (16-EI-0134), the Genetics of Inherited Eye Disease protocol (15-EI-0128), and the Pathogenesis and Genetics of Microphthalmia, Anophthalmia and Uveal Coloboma (MAC) protocol (13-EI-0049).

Offsite participants will be screened via phone or secure videoconference, and records will be requested for evaluation of affected participants. Both affected and unaffected eligible participants will undergo genetic counseling and will provide a blood sample and/or saliva sample for exome or genome sequencing. Biological relationships will be confirmed prior to exome or genome sequencing. Sequence data will be analyzed for primary variants and secondary findings, unless participants choose to opt-out of secondary analysis and reporting. All sequence variants deemed clinically relevant will be validated in a Clinical Laboratory Improvement Amendment (CLIA)-certified laboratory and the results will be returned to the participant in-person, secure videoconference, or by telephone.

Outcome Measures: This is an etiologic study that will generate molecular information about previously-recognized conditions for which participants did not have a molecular diagnosis, as well as molecular information for previously uncharacterized conditions involving the eye.

DETAILED DESCRIPTION:
Objective: The objective of this study is to identify genetic causes of inherited eye conditions through whole exome or whole genome sequencing (referred to as exome sequencing and genome sequencing in the remainder of the document). This includes identifying mutations in known genes or novel genes for recognized conditions, as well as identifying mutations in novel genes for previously uncharacterized genetic conditions involving the eye.

Study Population: We plan to recruit 1,685 participants, to include both participants with an eye condition under study and unaffected family members. Ideally unaffected family members will be parents of an affected participant.

Design: Participants will be self-referred or referred by an outside clinician. They will preferably be evaluated at the National Institutes of Health (NIH), but the option to participate offsite will be offered. Participants evaluated onsite will be recruited through other pre-existing NIH protocols, such as the National Eye Institute (NEI) Screening protocol (08-EI-0102), the NEI Ocular Natural History protocol (16-EI-0134), the Genetics of Inherited Eye Disease protocol (15-EI-0128), and the Pathogenesis and Genetics of Microphthalmia, Anophthalmia and Uveal Coloboma (MAC) protocol (13-EI-0049).

Offsite participants will be screened via phone or secure videoconference, and records will be requested for evaluation of affected participants. Both affected and unaffected eligible participants will undergo genetic counseling and will provide a blood sample and/or saliva sample for exome or genome sequencing. Biological relationships will be confirmed prior to exome or genome sequencing. Sequence data will be analyzed for primary variants and secondary findings, unless participants choose to opt-out of secondary analysis and reporting. All sequence variants deemed clinically relevant will be validated in a Clinical Laboratory Improvement Amendment (CLIA)-certified laboratory and the results will be returned to the participant in-person, secure videoconference, or by telephone.

Outcome Measures: This is an etiologic study that will generate molecular information about previously-recognized conditions for which participants did not have a molecular diagnosis, as well as molecular information for previously uncharacterized conditions involving the eye.

ELIGIBILITY:
* INCLUSION CRITERIA

To be eligible, participants must meet the following criteria:

1. Participant is affected with an eye condition under study or is a family member of an affected individual who will be informative for ES/GS analysis and interpretation.
2. Participant or legal guardian of participant understands and signs the informed consent document.

EXCLUSION CRITERIA

1. Participants who cannot comply with study procedures are ineligible.
2. Participants who are minors are ineligible if they do not have a parent/legal guardian who can consent and make decisions on their behalf. Participants who are or become decisionally impaired are ineligible if they do not have, or are unable to obtain, a legally authorized representative who can consent and make decisions on their behalf.
3. Participants who are minors and under joint custody are ineligible if parents disagree about study participation.
4. Prospective participants or their parent/legal guardians or legally authorized representatives who, based on the judgment of the team, appear to have impaired ability to understand and appropriately use complex medical and genetic information, or to cope with potentially life altering medical information, will be ineligible.

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study seeks to recruit patients with a diagnosis of inherited or congenital eye condition whose phenotype was confirmed either at the National Eye Institute (NEI) or through an outside clinician such as an ophthalmologist or geneticist. Select unaffected family members (in many cases, parents) will also be recruited in order to facilitate data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1685 (Estimated)
Dates: Start 2014-08-05 (Actual); Primary Completion 2029-08-05 (Estimated); Study Completion 2029-08-05 (Estimated)

PRIMARY OUTCOMES:
This is an etiologic study that will generate new genes or variants for inherited eye diseases. | Until the affected participant has received confirmed Primary Results (PRs). Unaffected family members may or may not receive any results, but their participation will be ongoing until their affected family member receives PRs.
  This is an etiologic study that will generate molecular information about previously-recognized conditions for which participants did not have a molecular diagnosis, as well as molecular information for previously uncharacterized eye conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Guan, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center,, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At this time, no IPD will be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-EI-0064.html